CLINICAL TRIAL: NCT02456935
Title: A Double-blind, Randomized, Active-controlled, Phase 3 Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Erosive Esophagitis
Brief Title: Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_301
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-12420 100 mg QD (Experimental): CJ-12420 100 mg, tablet, once daily, oral administration for up to 8 weeks
  Interventions: Drug: CJ-12420 100 mg QD
- Esomeprazole 40 mg QD (Active Comparator): Esomeprazole 40 mg, tablet, once daily, oral administration for up to 8 weeks
  Interventions: Drug: Esomeprazole 40 mg QD

INTERVENTIONS:
Drug: CJ-12420 100 mg QD — CJ-12420 100 mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose erosive esophagitis is not endoscopically healed at Week 4, subjects will receive additional 4 week treatment of CJ-12420 100 mg.
  Other Names: Not yet decided
  Arms: CJ-12420 100 mg QD
Drug: Esomeprazole 40 mg QD — Esomeprazole 40 mg tablets will be orally administered, once daily, for up to 8 weeks. For subjects whose erosive esophagitis is not endoscopically healed at Week 4, subjects will receive additional 4 week treatment of Esomeprazole 40 mg.
  Other Names: Nexium
  Arms: Esomeprazole 40 mg QD

SUMMARY:
The purpose of this study is to demonstrate the efficacy of CJ-12420, once daily (QD), compared to esomeprazole in patients with erosive esophagitis classified as Los Angeles (LA) classification grades A to D at Week 8

DETAILED DESCRIPTION:
This is a double blind, randomized, active controlled, phase 3 study. Subjects will be randomly assigned to one of the two treatment groups (CJ-12420 100 mg or esomeprazole 40 mg).

All subjects will be asked to take two tablets at the same time each day throughout the study, and also all subjects will be asked to record daytime and nighttime symptom in a subject diary on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 20 and 70 years
2. Subjects who had experienced heartburn and regurgitation within 7 days before visit 1. Entry into study also required that patients had experienced at least mild upper gastrointestinal symptoms on at least 2 days/week or at least moderate upper gastrointestinal symptoms on at least 1 day/week
3. Endoscopically confirmed erosive esophagitis as defined by LA Classification Grading System (A-D) within 14 days prior to randomization
4. Subjects who is able to understand and follow the instructions and is willing to participate throughout the entire study
5. Subjects who voluntarily signed written informed consent form
6. Subjects who agreed to use medically acceptable contraceptives during the period of study.

Exclusion Criteria:

1. Subjects who cannot undergo EGD
2. Subjects who have esophageal stenosis, ulcer stenosis, gastroesophageal varices, Barrett's esophagus, active gastric ulcer, gastrointestinal bleeding or malignant tumor confirmed by EGD
3. Subjects who have warning symptoms of malignant gastrointestinal tract such as odynophagia, severe dysphagia, bleeding, weight loss, anemia, or bloody stool
4. Subjects with eosinophilic esophagitis
5. Subjects diagnosed with primary esophageal motility disorder, IBS, IBD, etc. or with suspected IBS in the last 3 months
6. Subjects who have a history of gastric acid suppression surgery or upper gastrointestinal, esophageal surgery
7. Pregnant or lactating women
8. Subjects with a history of clinically significant hepatic, renal, cardiovascular, respiratory, endocrine and CNS system disorder
9. Subjects with a history of hypersensitivity to the active ingredient or excipients of the study drug, etc.
10. Subjects who participated in the other clinical trial within 4 weeks prior to randomization

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cumulative healing rate of erosive esophagitis at 8-week | 8 week

SECONDARY OUTCOMES:
Healing rate of erosive esophagitis at 4-week | 4 week
Symptom assessment by subject diary and questionnaire | 4 week or 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Chae Jung, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea